CLINICAL TRIAL: NCT05209529
Title: Neoadjuvant Olaparib and Durvalumab for Patients With BRCA-associated Triple Negative Breast Cancer
Brief Title: Chemo-free BRCA-targeted Neoadjuvant Strategy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn interest from grant provider
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1984-BCG; 2022-003594-33 (EudraCT Number)
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: TNBC - Triple-Negative Breast Cancer; BRCA1 Mutation; BRCA2 Mutation
Keywords: Olaparib; Durvalumab; PARPi
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — olaparib; durvalumab

STUDY DESIGN:
Intervention Model Description: Eligible patients after central screening are randomized to olaparib vs olaparib and durvalumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olaparib (Experimental): Olaparib treatment for a total of 16 weeks
  Interventions: Drug: olaparib
- Olaparib and durvalumab (Experimental): Olaparib and durvalumab treatment for a total of 16 weeks
  Interventions: Drug: olaparib; Drug: Durvalumab

INTERVENTIONS:
Drug: olaparib — olaparib 300 mg per os BID
Drug: Durvalumab — durvalumab 1500 mg IV Q4 weeks
  Arms: Olaparib and durvalumab

SUMMARY:
This is a multicenter randomized phase ll clinical trial to evaluate the pathological complete response (pCR) in the tumour burden (primary and lymph nodes) with olaparib alone or in the olaparib and durvalumab arm in TNBC patients candidate for neoadjuvant strategy showing a t/gBRCAmut or BRCAness/HRD profile.

DETAILED DESCRIPTION:
Eligible patients will be registered for central testing of BRCA mutatinal status and HRD/BRCAness profile with central review of ER, PgR, TILs and PD-L1.

Eligible patients will be randomly assigned to either olparib or olaparib and durvalumab (=neoadjuvant treatment) in a 1:1 ratio. The treatment duration in both arms will last 16 weeks and both treatments are considered as experimental treatments in this study.

After completion of neoadjuvant systemic treatment, patients will undergo surgery and followed-up for 2 years after investigational drug discontinuation. After surgery, adjuvant treatment will be left at the investigator's decision.

ELIGIBILITY:
Inclusion Criteria at registration:

* Histologically confirmed, invasive TNBC, defined as:

  * ER and PR negative (not eligible for endocrine therapy) defined as immunohistochemistry (IHC) nuclear staining ≤ 10% AND
  * HER2 negative (not eligible for anti-HER2 therapy):
* Early-stage disease, defined as cT1c-T2, N0-N1, M0
* Medically fit for a neoadjuvant strategy and for radical surgery as by the investigator's decision
* No prior systemic therapy nor definitive surgery for BC
* Age ≥18 years
* Women and men can be included
* ECOG performance status (PS) 0-1

Exclusion Criteria at registration:

* Previous treatment with a PARPi
* Previous treatment with an anti-PD-1/PD-L1, anti-PD-L2 or anti-CTLA-4 antibody
* Evidence of macroscopic distant metastases, investigated according to local institutional guidelines
* Patients who underwent sentinel node biopsy before neoadjuvant therapy
* History of previous invasive BC
* Bilateral and/or multifocal and/or multicentric BC
* Malabsorption syndrome or other chronic condition that would significantly interfere with enteral absorption
* History of allogenic transplantation of bone marrow or an organ.
* History of another primary malignancy.
* Myelodysplastic syndrome/acute myeloid leukaemia or features suggestive of such.
* Congenital long QT syndrome.
* History of active primary immunodeficiency

Inclusion criteria at randomization:

* Deleterious germline or somatic mutation in BRCA 1 and/or BRCA 2 or homologue repair deficiency (HRD) status as determined by central testing.
* Tumour tissue available from primary tumour (fine needle aspiration cytology or lymph node metastasis tissue are not acceptable).
* Normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

  * Haemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN
  * Total bilirubin ≤ 1.5 x ULN (exception: higher bilirubin in patients with confirmed Gilbert's syndrome are allowed according to the investigator's decision)
  * Creatinine clearance estimated of ≥ 51 mL/min/1.73m2 using the MDRD equation
* Body weight >30 kg
* Participation in translational research is mandatory
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test in the screening period and confirmed prior to treatment on day 1.
* Female patients of childbearing/reproductive potential must use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 3 months after the last dose of treatment. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Such methods include:

  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomized partner
  * Sexual abstinence (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient)
* Male patients must use a condom during treatment and for 3 months after the last dose of study treatment when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception (see above) if they are of childbearing potential.
* Female subjects who are breast feeding must discontinue nursing prior to the first dose of study treatment and until 3 months after the last study treatment.
* Registration to a National Health Care System

Exclusion criteria at randomization:

* Inability to swallow and/or retain oral tablets
* Blood transfusion within 28 days
* History of human immunodeficiency virus (HIV) (positive HIV 1/2-antibodies)
* Active Hepatitis B or Hepatitis C
* Active bacterial, viral, or fungal infection requiring systemic therapy
* History of active tuberculosis (TB, Bacillus Tuberculosis)
* History of idiopathic pulmonary fibrosis, drug-induced pneumonitis, organizing pneumonia, interstitial lung disease or evidence of active pneumonitis on screening (TAP-CT-scan)
* History of aortic disease (aneurysm or dissection)
* History of myasthenia gravis
* Mean QT interval corrected for heart rate (QTc) ≥ 500ms using Fridericia's Correction
* Uncontrolled intercurrent illness
* Psychiatric illness/social situations or addiction (chronic alcoholism or drug addiction) that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* Any other serious or uncontrolled illness or abnormality that, in the judgment of the investigator, limits compliance with study requirement, substantially increases risk of incurring AEs or compromises the ability to give written informed consent.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study treatment.
* Any concurrent systemic chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment.
* Any unresolved toxicity (Common Terminology Criteria for Adverse Event (CTCAE) grade ≥ 2) caused by previous cancer therapy, excluding alopecia, vitiligo.

  * Patients with Grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with olaparib and/or durvalumab may be included only after consultation with the study physician.
* Concomitant use of strong CYP3A inhibitors.The required washout period prior to starting study treatment (olaparib) is 2 weeks.
* Concomitant use of strong CYP3A inducers. The required washout period prior to starting study treatment (olaparib) is 5 weeks for phenobarbital and 3 weeks for other agents.
* Major surgery within 4 weeks prior to the first dose of study treatment. Patients must have recovered from the surgical procedure. Implanted port placement is not considered as a major surgery.
* Known allergy or hypersensitivity to olaparib or durvalumab, or to any excipient.
* Contraindication to MRI or to the contrast medium used for MRI (gadolinium).
* Participation in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Female patients who are pregnant or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 3 months after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2028-09-06 (Estimated); Study Completion 2030-07-18 (Estimated)

PRIMARY OUTCOMES:
rate of pathological complete response (pCR) at the time of surgery | 5 years from first patient in
  pCR is defined as the absence of invasive residual disease in the breast and in the axillary lymph nodes (ypT0/is ypN0).

SECONDARY OUTCOMES:
2-year overall survival (OS) rate | 7.5 years from first patient in
  OS is defined as date of randomization to the date of death, whatever comes first
Other pathological response | 7.5 years from first patient in
  Residual cancer burden score (RCB), defined on the specimen collected at the time of surgery
Probability of being event-free at 2 years | 7.5 years from first patient in
  events considered being disease progression on neoadjuvant therapy, any event precluding surgery, locoregional recurrence, distant recurrence, second primary invasive cancer (breast and non-breast origin) and death from any cause
Surgery rate | 7.5 years from first patient in
Breast conservation rate | 7.5 years from first patient in
Treatment response rate according to RECIST v1.1 | 7.5 years from first patient in
Safety | 7.5 years from first patient in
  Rate of Adverse events not related directly with the surgical procedure (NCI-CTCAE Version 5.0) Rate of Post-operative complications (Clavien-Dindo Classification of Surgical Complications)
Global health status/QoL score | 7.5 years from first patient in
  score according to EORTC QLQ-C30 questionnaire
Score on the Systemic side effects scale | 7.5 years from first patient in
  according to the modified QLQ-BR45 (IL170) questionnaire

OTHER OUTCOMES:
Exploratory endpoints: the impact of olaparib alone or olaparib in combination with durvalumab on ovarian function (in patients ≤ 50 years) | 7.5 years from first patient in
  Change in ovarian reserve over time as measured by AMH; Proportion of premenopausal women at baseline who become postmenopausal after neoadjuvant treatment and during follow-up as measured by FSH and E2
Exploratory endpoints: Translational research | 7.5 years from first patient in
  Preliminary assessment of biomarkers that might act as pharmacodynamic indicators and predictors of activity of the experimental treatment by IHC, immunomonitoring, genetic and imaging studies.
Exploratory endpoints: To assess the evolution of the other scales HRQoL in both arms | 7.5 years from first patient in
  according to EORTC QLQ-C30 questionnaire and the modified QLQ-BR45 (IL170) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Brain, Study Chair — Institut Curie Paris

IPD SHARING:
Plan to Share IPD: No